CLINICAL TRIAL: NCT05913687
Title: Automated Imaging Differentiation of Parkinsonism
Acronym: AIDP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Augusta University (Other); Albany Medical College (Other); Beth Israel Deaconess Medical Center (Other); Duke University (Other); Johns Hopkins University (Other); Massachusetts General Hospital (Other); Northwestern University (Other); Ottawa Hospital Research Institute (Other); Penn State University (Other); University of Alabama at Birmingham (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of Chicago (Other); University of Michigan (Other); University of Minnesota (Other); University of South Florida (Other); Centre for Addiction and Mental Health (Other); Wake Forest University (Other); Washington University School of Medicine (Other); University of Kentucky (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202002350; PRO00028349 (Other: UF); 5U01NS119562 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Multiple System Atrophy, Parkinson Variant; Progressive Supranuclear Palsy
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's disease: Clinically diagnosed Parkinson's disease
  Interventions: Diagnostic Test: AIDP
- Multiple System Atrophy, Parkinsonian variant: Clinically diagnosed Multiple System Atrophy, Parkinsonian variant
  Interventions: Diagnostic Test: AIDP
- Progressive Supranuclear Palsy: Clinically diagnosed Progressive Supranuclear Palsy
  Interventions: Diagnostic Test: AIDP

INTERVENTIONS:
Diagnostic Test: AIDP — Machine learning algorithm of imaging data

SUMMARY:
The purpose of this study is to test the performance of the AID-P across 21 sites in the Parkinson Study Group. Each site will perform imaging, clinical scales, diagnosis, and will upload the data to the web-based software tool. The clinical diagnosis will be blinded to the diagnostic algorithm and the imaging diagnosis will be compared to the movement disorders trained neurologist diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis within 5-9 years of baseline date
* MSAp diagnosis
* PSP diagnosis

Exclusion Criteria:

* metal implants in the body that preclude an MRI (pacemaker, metallic clip, neurostimulator, etc)
* claustrophobia
* pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 40 and 80 who meet one of the three diagnoses: PD, MSAp, or PSP
  *As of 11/9/23, we have filled the cohorts for both PD and PSP patients. We are only enrolling MSAp patients at this time.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Predicted diagnosis accuracy | 12-18 months
  utilizing the automated imaging differentiation of Parkinsonism (AIDP) tool to predict diagnosis compared to the expertise of two movement disorder specialists

CONTACTS AND LOCATIONS:
Locations (21):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Pennsylvania State University, Hershey, Pennsylvania
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa
  - Centre for Addiction and Mental Health, Toronto

IPD SHARING:
Plan to Share IPD: No